CLINICAL TRIAL: NCT00319514
Title: Randomized Phase II Trial of Two Different Schedules of Docetaxel Plus Cisplatin as First-Line Therapy in Advanced Non-Small Cell Lung Cancer
Brief Title: Weekly Versus 3-Weekly Docetaxel Plus Cisplatin for Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMO-LU-42
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
To evaluate the toxicity and efficacy of docetaxel and cisplatin combination on two schedules in patients with previously untreated, advanced NSCLC.

DETAILED DESCRIPTION:
The combination of docetaxel 75 mg/m2 and cisplatin 60-80 mg/m2 administered every 3 weeks is one of the most commonly used chemotherapy regimen in Korea for the first-line treatment of advanced NSCLC. Although the 3-weekly regimen is active and tolerated, it is associated with a significant incidence of severe neutropenia, often complicated by fever. Therefore, there has been increasing interest in the use of a weekly administration of docetaxel as a way of reducing its hematologic toxicity. We designed this randomized phase II trial to evaluate the safety profile and antitumor activity of two different schedules of docetaxel plus cisplatin given as first-line therapy in patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven non-small cell lung cancer
* no prior chemotherapy or only adjuvant chemotherapy which had been completed >6 months before registration
* ECOG performance status 0 to 2
* measurable lesion(s)
* normal marrow, hepatic and renal functions
* provision of written informed consent

Exclusion Criteria:

* active infection or severe comorbidities
* history of anaphylaxis of any origin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Start 2004-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea